CLINICAL TRIAL: NCT05101798
Title: The Role of 5-Aminolevulinic Acid Fluorescence-Guided Surgery in Head and Neck Cancers: a Pilot Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: NX Development Corporation closed the trial
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: NX Development Corp (Industry)
Responsible Party: Principal Investigator, Alfred-Marc Iloreta, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-20-00713
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Neoplasm; Skull Base Neoplasm
Keywords: head and neck tumor; skull base tumor; neoplasm
MeSH Terms: conditions — Neoplasms; Skull Base Neoplasms; Head and Neck Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5-aminolevulinic acid hydrochloride (Gleolan®) (Experimental): Gleolan® is available in colorless glass vials containing 1.5 g 5-aminolevulinic acid hydrochloride (Gleolan®) Gleolan® is administered orally to patients prior to tumor removal by surgery (20 mg/kg BW).
  Interventions: Drug: 5-Aminolevulinic acid Hydrochloride

INTERVENTIONS:
Drug: 5-Aminolevulinic acid Hydrochloride — The closure consists of colorless glass vial (Type II, Ph Eur) and bromobutyl-rubber stopper ø 20 mm (Type I, Ph Eur) and flip cap. The powder for oral solution is intended for single (partial) use. To prepare the ready-to-use solution the content of one vial is dissolved in 50 ml of water or apple juice. The concentration of the reconstituted solution is 3%. Gleolan® is administered orally to patients prior to tumor removal by surgery (20 mg/kg BW). The reconstituted solution may be prepared up to 24 hours prior to use if protected from light. It should be given 3 hours (range 3-5 hours) prior to planned induction of anesthesia for surgery, although its effect is present for up to 8-12 hours. This step is critical for an optimal visualization of tumor tissue due to pharmacokinetic properties of Gleolan®.
  Other Names: Gleolan®

SUMMARY:
This study allows head and neck cancer surgeons to specifically visualize cancerous cells apart from normal healthy tissue. 5-aminolevulinic acid (5-ALA) is a safe and effective FDA-approved agent successfully used by neurosurgeons for FGS of different brain tumors is given to the patients preoperatively. Using specific wavelengths of light as well as specialized magnified lenses the surgeons use this technique to assist in tumor resection.

DETAILED DESCRIPTION:
Treatment for many head and neck cancer involves surgical resection, or removal, of the tumor. A potential outcome of surgery is subtotal resection, in which some cancerous material fails to be removed resulting in tumor recurrence and lower overall survival. Achieving total resection without interfering with normal tissue is a challenge due the critical anatomical structures of the head and neck. Fluorescent-guided surgery (FGS) is a new method of intraoperative imaging that can be used to clearly visualize cancerous tissue aprt from normal tissue during surgery in real-time. Before surgery, an agent that preferentially enters tumor cells is given to the patient. Tumor cells then glow brightly when exposed to specific wavelengths of light during surgery, allowing the surgeon to easily distinguish between healthy and cancerous tissue. 5-aminolevulinic acid (5-ALA) is a safe and effective FDA approved agent successfully used by neurosurgeons for FGS of different brain tumors which has not been assessed for use in head and neck cancers. The aim of the study is to determine if 5-ALA can be effectively used in FGS for different types of head and neck cancers, and if it will improve survival, tumor regrowth, and other outcomes for patients. 23 patients will be enrolled from the Mount Sinai Hospital, New York Eye and Ear Infirmary and Mount Sinai Union Square Faculty Practices over a 1 year period and will be completed by December 2022.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in this trial must have had documentation of a new or recurrent head and neck or skull base tumor for which surgical resection is indicated and has been planned. These patients will include those with newly diagnosed or recurrent malignancies.
* Age 18-80
* Karnofsky score >60%
* Subjects must have normal organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcl
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR Creatinine clearance >60 mL/min/1.73m2 for patients with creatinine levels above institutional normal as defined per institution.
* The effects of Gleolan® (5-ALA) on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. A pregnancy test will be performed for all women of childbearing ability prior to surgery (see Exclusion Criteria below). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.
* all upper aerodigestive head and neck cancers

Exclusion Criteria:

* Patients with non-resectable tumors or not deemed surgical candidates
* History of allergic reactions attributed to compounds of similar chemical/biologic composition to ALA.
* Personal or family history of porphyria
* Uncontrolled concurrent illness including but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness//social situations that would limit compliance with study requirements
* Women who are pregnant or become pregnant will be excluded from the trial as it is unknown if ALA is teratogenic or has abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 5-ALA breastfeeding should be discontinued if the mother is treated with 5-ALA.
* Prior history of GI perforation, diverticulitis, and or/peptic ulcer disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred-Marc Iloreta, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mount Sinai Union Square, New York, New York
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
Data will be de-identified and aggregated in all reporting

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was opened on 9/14/2021 and study was actively recruiting through Jan 14, 2025. The date of the last study visit was Dec 25, 2022. On Jan 14, 2025, the sponsor contacted the study team regarding closing the study. The study was officially closed on Feb 25, 2025.
Period: Overall Study
Arm/Group | 5-aminolevulinic Acid Hydrochloride (Gleolan®)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 5-aminolevulinic Acid Hydrochloride (Gleolan®)
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 60 [33 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Test Result of PPIX Tissue Fluorescence
Description: The feasibility of using oral Gleolan® as an adjunct diagnostic imaging tool for malignant tumor tissue fluorescence will be primarily assessed by computing sensitivity of intraoperative Gleolan® induced PPIX tissue fluorescence.
  PPIX tissue fluorescence will be defined categorically as "no" (score 0), "low" (score 1), "medium" (score 2), and "high" (score 3) by operative surgeon, and images will be recorded. For purposes of computing measures of diagnostic performance a score of 0 will be considered a negative test result and a score of 1, 2 or 3 will be considered a positive test result.
Time Frame: Through completion of surgery, up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 5-aminolevulinic Acid Hydrochloride (Gleolan®)
Number analyzed (Participants) | 7
Participants
  0 | 1
  1 | 0
  2 | 0
  3 | 6

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | 5-aminolevulinic Acid Hydrochloride (Gleolan®)
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-aminolevulinic Acid Hydrochloride (Gleolan®) (N=7)
Mild photosensitivity reaction (CTCAE grade I) (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
The renewal arm of the study (2022-2025) depended on materials from NX Development Corporation (Aladuck endoscope and Gleolan (5-ALA) drug). Thus, when NX Development Corporation decided to close the study, the researchers were unable to continue study activities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT05101798/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT05101798/ICF_001.pdf